CLINICAL TRIAL: NCT03096795
Title: Safety, Tolerability, Pharmacokinetics and Immunogenicity of MEDI3506 Administered as Single Ascending Doses in Healthy Adult Subjects, as Multiple Ascending Doses in COPD Subjects and Single Dose in Healthy Japanese Subjects
Brief Title: Safety and Tolerability of MEDI3506 in Healthy Participants, in Participants With COPD and Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D9180C00001
Record Dates: First submitted 2017-03-01; First posted 2017-03-30 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Part I (SAD) - Healthy Participants; Part II (MAD) - Chronic Obstructive Pulmonary Disease; Part III (J-SD) - Healthy Japanese Participants
Keywords: MEDI3506; Safety; Tolerability; Pharmacokinetics; Immunogenicity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Part 1: Placebo (Placebo Comparator): Healthy participants with a history of mild atopy and proven sensitivity to house dust mite (HDM) will receive a single dose of placebo matched to MEDI3506 subcutaneously or intravenously.
  Interventions: Drug: MEDI3506; Drug: Placebo
- Part 1: MEDI3506 SC Dose 1 (Experimental): Healthy participants with a history of mild atopy and proven sensitivity to HDM will receive a single MEDI3506 Dose 1 subcutaneously.
  Interventions: Drug: MEDI3506
- Part 1: MEDI3506 SC Dose 2 (Experimental): Healthy participants with a history of mild atopy and proven sensitivity to HDM will receive a single MEDI3506 Dose 2 subcutaneously.
  Interventions: Drug: MEDI3506
- Part 1: MEDI3506 SC Dose 3 (Experimental): Healthy participants with a history of mild atopy and proven sensitivity to HDM will receive a single MEDI3506 Dose 3 subcutaneously.
  Interventions: Drug: MEDI3506
- Part 1: MEDI3506 SC Dose 4 (Experimental): Healthy participants with a history of mild atopy and proven sensitivity to HDM will receive a single MEDI3506 Dose 4 subcutaneously.
  Interventions: Drug: MEDI3506
- Part 1: MEDI3506 SC Dose 5 (Experimental): Healthy participants with a history of mild atopy and proven sensitivity to HDM will receive a single MEDI3506 Dose 5 subcutaneously.
  Interventions: Drug: MEDI3506
- Part 1: MEDI3506 SC Dose 6 (Experimental): Healthy participants with a history of mild atopy and proven sensitivity to HDM will receive a single MEDI3506 Dose 6 subcutaneously.
  Interventions: Drug: MEDI3506
- Part 1: MEDI3506 IV Dose 6 (Experimental): Healthy participants with a history of mild atopy and proven sensitivity to HDM will receive a single MEDI3506 Dose 6 intravenously.
  Interventions: Drug: MEDI3506
- Part 2: Placebo (Placebo Comparator): Participants with COPD will receive 3 administration of placebo matched to MEDI3506 subcutaneously two weeks apart over a 4-week dosing period (doses on Days 1, 15, and 29).
  Interventions: Drug: MEDI3506; Drug: Placebo
- Part 2: MEDI3506 SC Dose 4 (Experimental): Participants with COPD will receive 3 administration of MEDI3506 Dose 4 subcutaneously two weeks apart over a 4-week dosing period (doses on Days 1, 15, and 29).
  Interventions: Drug: MEDI3506
- Part 2: MEDI3506 SC Dose 5 (Experimental): Participants with COPD will receive 3 administration of MEDI3506 Dose 5 subcutaneously two weeks apart over a 4-week dosing period (doses on Days 1, 15, and 29).
  Interventions: Drug: MEDI3506
- Part 2: MEDI3506 SC Dose 6 (Experimental): Participants with COPD will receive 3 administration of MEDI3506 Dose 6 subcutaneously two weeks apart over a 4-week dosing period (doses on Days 1, 15, and 29).
  Interventions: Drug: MEDI3506
- Part 3: Placebo (Placebo Comparator): Healthy Japanese participants will receive a single dose of placebo matched to MEDI3506 intravenously.
  Interventions: Drug: MEDI3506; Drug: Placebo
- Part 3: MEDI3506 IV Dose 6 (Experimental): Healthy Japanese participants will receive a single MEDI3506 Dose 6 intravenously.
  Interventions: Drug: MEDI3506

INTERVENTIONS:
Drug: MEDI3506 — Healthy participants with a history of mild atopy and proven sensitivity to HDM will receive a single MEDI3506 Dose 1 or Dose 2 or Dose 3 or Dose 4 or Dose 5 or Dose 6 subcutaneously and Dose 6 intravenously in Part 1. Participants with COPD will receive 3 administration of MEDI3506 Dose 4 or Dose 5 or Dose 6 subcutaneously two weeks apart over a 4-week dosing period in Part 2. Healthy Japanese participants will receive a single dose of MEDI3506 Dose 6 intravenously in Part 3.
Drug: Placebo — Healthy participants with a history of mild atopy and proven sensitivity to HDM will receive a single dose of placebo matched to MEDI3506 subcutaneously or intravenously in Part 1. Participants with COPD will receive 3 administration of placebo matched to MEDI3506 subcutaneously two weeks apart over a 4-week dosing period in Part 2. Healthy Japanese participants will receive a single dose of placebo matched to MEDI3506 intravenously in Part 3.
  Arms: Part 1: Placebo; Part 2: Placebo; Part 3: Placebo

SUMMARY:
This is a Phase 1, randomised, blinded, placebo controlled, study designed to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity response to single and multiple doses of MEDI3506.

DETAILED DESCRIPTION:
This is a Phase 1, randomised, blinded, placebo controlled, study designed to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity response to single and multiple doses of MEDI3506 administered by either subcutaneous (SC) or intravenous (IV) routes.

Part I: Single Ascending Doses in Healthy Participants with a History of Mild Atopy

Part II: Multiple Ascending Doses in Participants with Global Initiative for Chronic Obstructive Lung Disease (GOLD) I-II Chronic Obstructive Pulmonary Disease (COPD)

Part III: Single Dose in Healthy Japanese Participants

ELIGIBILITY:
Inclusion Criteria Part 1

1. Healthy volunteers aged 18 through 55 years at the time of consent.
2. Non-smokers, healthy current smokers, and ex-smokers are permitted.
3. Pre-bronchodilator forced expiratory volume in 1 second (FEV1) >= 80% predicted (using the Global Lung Initiative [GLI] predicted values) at screening.
4. Body mass index (BMI) of 19.0 through 32.0 kg/m^2 at screening.
5. Current history of mild atopy.

Inclusion Criteria Part 2

1. Aged 40 through 80 years at the time of screening.
2. BMI of 19.0 through 35.0 kg/m^2 at screening.
3. Participants must be current on pneumococcus and annual influenza vaccines.
4. Documented history of COPD with a post-bronchodilator FEV1/force vital capacity (FVC) <0.70 and a post-bronchodilator FEV1 ≥50% predicted at screening.
5. Clinically stable and free from an acute exacerbation of COPD for 8 weeks prior to Day 1.
6. Current or ex-smoker with a tobacco history of ≥10 pack-years.

Inclusion Criteria Part 3

1. Japanese participants must have been born in Japan, have both parents and grandparents of Japanese origin, and not have lived outside of Japan for more than 5 years.
2. Healthy participants aged 20 through 55 years at the time of consent.
3. Non-smokers, healthy current smokers, and ex-smokers are permitted.
4. BMI of 18.0 through 32.0 kg/m^2 at screening.

Exclusion Criteria Part 1

1. Concurrent enrollment in another clinical study involving a study treatment.
2. Received administration of study drug or participated in a device trial within 3 months, prior to screening (Visit 1).
3. Participant is a participating investigator, sub-investigator, study coordinator or employee of the participating site, or is a first-degree relative of the aforementioned.
4. Any active medical or psychiatric condition or other reason which, in the opinion of the investigator or medical monitor, may compromise the safety of the participant in the study or interfere with evaluation of the investigational product or reduce the participant's ability to participate in the study.
5. Any clinically relevant abnormal findings on physical examination of the cardiovascular system including electrocardiogram (ECG) and vital signs at screening or randomization.
6. Abnormal vital signs, after 10 minutes supine rest.

Exclusion Criteria Part 2

1. Concurrent enrolment in another clinical study involving investigational treatment.
2. Received administration of study drug or participated in a device trial within 3 months, prior to screening (Visit 1).
3. Participant is a participating investigator, sub-investigator, study coordinator, or employee of the participating site, or is a first-degree relative of the aforementioned.
4. Any active medical or psychiatric condition or other reason that, in the opinion of the investigator, would interfere with evaluation of the study drug or interpretation of participant's safety or study results. This includes, but is not limited to:

   * Uncontrolled diabetes
   * Hypertension during the screening period
   * Significant or unstable ischaemic heart disease, arrhythmia, cardiomyopathy, heart failure
   * Clinically significant Aortic stenosis
   * Pulmonary Arterial Hypertension

Exclusion Criteria Part 3

1. Concurrent enrolment in another clinical study involving study treatment.
2. Received administration of study drug or participated in a device trial within 3 months, prior to screening (Visit 1).
3. Any active medical or psychiatric condition or other reason which, in the opinion of the investigator or medical monitor, may compromise the safety of the participant in the study or interfere with evaluation of the study product or reduce the participant's ability to participate in the study.
4. Any clinically relevant abnormal findings on physical examination of the cardiovascular system including ECG and vital signs at screening, and Day 1(pre-dose).
5. Any other clinically relevant abnormal findings on physical examination or laboratory testing including hematology, coagulation, clinical chemistry or urinalysis at screening or randomisation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs), and Treatment-emergent Adverse Events of Special Interest (TEAESI) in Part 1, Part 2, and Part 3 | From Day 1 through Day 169
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. An adverse event of special interest (AESI) was defined as any serious or nonserious event of scientific and medical interest specific to understand the study drug.
Number of Participants With Grade 2 or More Toxicity Grades Reported in Laboratory Parameters at Day 169 for Part 1, Part 2, and Part 3 | Day 169
  Number of participants with Grade 2 or more toxicity grades reported in laboratory parameters are reported. Abnormal clinical laboratory parameters defined as any abnormal finding during analysis of hematology and serum chemistry.
Changes From Baseline in Blood Pressure at Day 169 in Part 1, Part 2, and Part 3 | Day 169
  Change from baseline in blood pressure at Day 169 in Part 1, Part 2, and Part 3 are reported.
Changes From Baseline in Pulse Rate at Day 169 in Part 1, Part 2, and Part 3 | Baseline (Day 1) and Day 169
  Change from baseline in pulse rate at Day 169 in Part 1, Part 2, and Part 3 is reported.
Changes From Baseline in Respiratory Rate at Day 169 in Part 1, Part 2, and Part 3 | Baseline (Day 1) and Day 169
  Change from baseline in respiratory rate at Day 169 in Part 1, Part 2, and Part 3 are reported.
Changes From Baseline in Body Temperature Rate at Day 169 in Part 1, Part 2, and Part 3 | Baseline (Day 1) and Day 169
  Change from baseline in body temperature at Day 169 in Part 1, Part 2, and Part 3 are reported.
Number of Participants With Change From Baseline in QTcF in Part 1, Part 2, and Part 3 | Baseline (Day 1) and Day 169
  Number of participants with change from basleine in QTcF in Part 1, Part 2, and Part 3 are reported. The change from baseline in QTcF at Day 169 data are reported in 3 categories as: <= 30 msec, > 30 to <= 60 msec, and > 60 msec.

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) of MEDI3506 After Single Dose for Part 1 and Part 3 | Day 1 (predose for all arms; except predose and end of infusion for MEDI3506 IV Dose 6 arms), Day 2, Day 3, Day 4, Day 5, Day 8, Day 15, Day 29, Day 43, Day 57, Day 85, Day 113, Day 141, and Day 169
  The Cmax of MEDI3506 after single dose for Part 1 and Part 3 are reported.
Time to Maximum Concentration (Tmax) of MEDI3506 After Single Dose for Part 1 and Part 3 | Day 1 (predose for all arms; except predose and end of infusion for MEDI3506 IV Dose 6 arms), Day 2, Day 3, Day 4, Day 5, Day 8, Day 15, Day 29, Day 43, Day 57, Day 85, Day 113, Day 141, and Day 169
  The Tmax of MEDI3506 after single dose for Part 1 and Part 3 is reported.
Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of MEDI3506 After Single Dose for Part 1 and Part 3 | Day 1 (predose for all arms; except predose and end of infusion for MEDI3506 IV Dose 6 arms), Day 2, Day 3, Day 4, Day 5, Day 8, Day 15, Day 29, Day 43, Day 57, Day 85, Day 113, Day 141, and Day 169
  The AUC0-inf of MEDI3506 after single dose for Part 1 and Part 3 are reported.
Terminal Elimination Half-life (t1/2) of MEDI3506 After Single Dose for Part 1 and Part 3 | Day 1 (predose for all arms; except predose and end of infusion for MEDI3506 IV Dose 6 arms), Day 2, Day 3, Day 4, Day 5, Day 8, Day 15, Day 29, Day 43, Day 57, Day 85, Day 113, Day 141, and Day 169
  The t1/2 of MEDI3506 after single dose for Part 1 and Part 3 are reported.
Apparent Clearance (CL/F) of MEDI3506 From Body After Single Dose for Part 1 and Part 3 | Day 1 (predose for all arms; except predose and end of infusion for MEDI3506 IV Dose 6 arms), Day 2, Day 3, Day 4, Day 5, Day 8, Day 15, Day 29, Day 43, Day 57, Day 85, Day 113, Day 141, and Day 169
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Total clearance from the body (CL) from Part 1 and Part 3 after intravenous administration or apparent systemic clearance (CL/F) after subcutaneous administration in Part 1 of the study are reported.
Trough Serum Concentration (Ctrough) of MEDI3506 After 1st Dose in Part 2 | Day 1 (predose), Day 3, Day 8, Day 15 (predose)
  Lowest serum concentration of MEDI3506 observed within the dosing interval after 1st dose in Part 2 is reported.
Trough Serum Concentration (Ctrough) of MEDI3506 After 3rd Dose in Part 2 | Day 29 (predose), Day 36, and Day 43
  Lowest serum concentration of MEDI3506 observed within the dosing interval after 3rd dose in Part 2 is reported.
Terminal Elimination Half-life (t1/2) of MEDI3506 in Part 2 | Day 36, Day 43, Day 57, Day 85, Day 113, Day 141, and Day 169
  The t1/2 of MEDI3506 after 3rd dose in Part 2 is reported.
Number of Participants With Positive Anti-drug Antibodies (ADA) to MEDI3506 treatment in Part 1, Part 2, and Part 3 | Part 1 and Part 3: Day 1 (predose), Day 29, Day 57, Day 85, Day 113, Day 141, and Day 169; Part 2: Day 1 (predose), Day 29, Day 85, and Day 169
  Number of participants with positive ADA to MEDI3506 treatment after single administration of MEDI3506 (Part 1 and Part 3) and after multiple dose administration of MEDI3506 (Part 2) at any time point during the study are reported.

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MBChB, FFPM. MSc, Principal Investigator — Parexel; David Singh, MD, Principal Investigator — Medicines Evaluation Unit
Locations (2):
- United Kingdom (2):
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search